CLINICAL TRIAL: NCT02180555
Title: Incidence and Predisposing Factors for the Development of Glucose Metabolism Disturbances and Diabetes Mellitus After Intensive Care Admission
Brief Title: Diabetes Mellitus After Intensive Care Admission
Acronym: DIAFIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Christophe De Block (Other)
Responsible Party: Sponsor-Investigator, Christophe De Block, MD, PhD, University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Other Study IDs: EC 12/2/22; B300201213039 (Other: Belgisch registratienummer)
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Stress Hyperglycemia; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ICU patients
  Interventions: Other: Oral glucose tolerance test

INTERVENTIONS:
Other: Oral glucose tolerance test

SUMMARY:
Stress hyperglycaemia is commonly observed during hospitalization in the intensive care unit (ICU) and has been shown to adversely influence outcome. It has been hypothesized that, when it occurs in previously non-diabetic patients, it reflects a latent disturbance of the glucose metabolism. Assessing the incidence of this phenomenon and identifying its risk factors could support prevention, detection and early treatment of impending diabetes mellitus type 2. We will perform a glucose tolerance test approximately 6-9 months post-ICU admission to screen for disorders of glucose metabolism. Furthermore, we examined characteristics that could have predicted the post-discharge disturbances: patient characteristics, parameters of disease severity and of glucose metabolism, as well as the FINDRISC (Finnish Diabetes Risc Score). We plan to enroll 400 patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old)
* admitted for 36 hours or longer to the ICU
* still alive 6 months after ICU discharge

Exclusion Criteria:

* known Diabetes Mellitus or any other glucose tolerance disturbance
* an estimated short life expectancy
* pregnancy
* a history of transplantation or acute pancreatic disease
* language barrier preventing a clear understanding of the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Glucose metabolism disturbance | 6-9 months after ICU discharge
  At a follow-up visit, patients will have their blood glucose levels sampled both after fasting and 2 hours after an oral glucose tolerance test (OGTT). HbA1c levels will be sampled once as well. Possible disturbances in glucose metabolism are the following: isolated impaired fasting glucose (IFG) = fasting plasma glucose (FPG) level of 100-125 mg/dl with the 2-h value after OGTT <140 mg/dl. Isolated impaired glucose tolerance (IGT) = 2-h value after OGTT of 140-199 mg/dl with the fasting level <100 mg/dl. Patients with combined characteristics of IFG and IGT fulfill both criteria (FPG = 100-125 mg/dl and 2-h value after OGTT = 140-199 mg/d). Diabetes mellitus is diagnosed when a patient has one of the following criteria: FPG more or equal to 126mg/dl, 2-h value after OGTT more or equal to 200 mg/dl, HbA1c more or equal to 6.5%.

SECONDARY OUTCOMES:
Patient characteristics predicting adverse outcome | 6-9 months after ICU discharge
  We will assess the effect of the patient's length, weight, body mass index (BMI), reason for admission, preadmission home medication, treatment during admission (steroids, vasopressors, inotropics, mechanical ventilation, insulin, total parenteral nutrition (TPN), laboratory values including blood glucose and HbA1c on intensive care unit (ICU) admission on our primary outcome parameter. Moreover, we will take into account the Simplified Acute Physiology Score (SAPS-3) and the daily Sequential Organ Failure Assessment (SOFA) score as parameters for disease severity, together with vasopressor or inotropic therapy, mechanical ventilation and length of stay at the hospital and ICU. Furthermore, our patients will complete the Finnish Diabetes Risk Score (FINDRISC) questionnaire during their follow-up visit, and we will compare this result with the primary outcome parameter as well.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerpen, Belgium

REFERENCES:
- [Background] Gornik I, Vujaklija-Brajkovic A, Renar IP, Gasparovic V. A prospective observational study of the relationship of critical illness associated hyperglycaemia in medical ICU patients and subsequent development of type 2 diabetes. Crit Care. 2010;14(4):R130. doi: 10.1186/cc9101. Epub 2010 Jul 8. PMID 20615210
- [Derived] Van Ackerbroeck S, Schepens T, Janssens K, Jorens PG, Verbrugghe W, Collet S, Van Hoof V, Van Gaal L, De Block C. Incidence and predisposing factors for the development of disturbed glucose metabolism and DIabetes mellitus AFter Intensive Care admission: the DIAFIC study. Crit Care. 2015 Oct 2;19:355. doi: 10.1186/s13054-015-1064-9. PMID 26428846